CLINICAL TRIAL: NCT03687931
Title: A Phase 1/2 Dose-Ranging, Open-Label, Randomized, Clinical Study to Assess the Efficacy and Safety of Dexamethasone Ophthalmic Suspension Eye Drops for the Treatment of Inflammation Associated With Cataract Surgery
Brief Title: A Clinical Study to Assess the Efficacy and Safety of Dexamethasone Suspension for Cataract Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: iDrop, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-01
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Inflammation Eye
MeSH Terms: conditions — Endophthalmitis | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Dexamethasone suspension dose level 1
  Interventions: Drug: Dexamethasone
- Arm 2 (Experimental): Dexamethasone suspension dose level 2
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Drop

SUMMARY:
Patients at least 40 years of age who are undergoing cataract surgery will be randomized to receive treatment with one of two dose levels of dexamethasone ophthalmic suspension eye drops to determine if the drops decrease inflammation inside the eye and are safe after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 40 years of age scheduled for unilateral cataract surgery by phacoemulsification with posterior chamber intraocular lens implantation.

Exclusion Criteria:

* Patients who have received a periocular corticosteroid injection in the study eye in the 3 months prior to screening.
* Patients who anticipate requiring treatment with any corticosteroids by any route, except inhalation, during the study.
* Patients who are known steroid responders

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-26 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Anterior Chamber Cell | 30 days
  Number of cells in the anterior chamber

CONTACTS AND LOCATIONS:
Overall Officials: William White, Study Chair — iDrop, Inc.
Locations (1):
- Arizona Eye Center, Chandler, Arizona, United States